CLINICAL TRIAL: NCT06679114
Title: Preventing Mental Disorders Among Women Internally Displaced by War in Ukraine: The SHAWL Trial
Acronym: SHAWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-45281; R34MH134077 (NIH)
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Mental Health Disorder; War-Related Trauma; Acceptance and Commitment Therapy; Depressive Symptoms Mild to Moderate in Severity; Refugee Health; Prevention
Keywords: Displacement; Women's health; Ukraine
MeSH Terms: conditions — Anxiety Disorders; Mental Disorders; War-Related Injuries | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: ACT Therapy (Experimental): Participants randomized to this group will receive a single-session ACT intervention
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Attention control (Active Comparator): Participants in the control group will receive minimally enhanced usual care to receive treatment as usual enhanced by a health information group session.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The single-session ACT group intervention will involve a mixture of didactic instruction, discussion, metaphors, and experiential activities. ACT activities will help women notice and accept that negative thoughts, emotions, and experiences while being displaced by war are part of migratory and post-migratory life. ACT activities will also help them identify, reorient towards, and commit to values-consistent behaviors through effective goal-setting. The single-session will be approximately 3 hours long.
  Arms: Behavioral: ACT Therapy
Behavioral: Attention control — Usual care will be minimally enhanced by providing participants with an educational information session that provides information on health promotion.
  Arms: Attention control

SUMMARY:
This study is a randomized controlled trial among 120 recently displaced women to determine the effectiveness of a single-session Acceptance and Commitment Therapy (ACT) group therapy on prevention of development of mental health disorders or worsened mental health symptoms.

DETAILED DESCRIPTION:
The war in Ukraine has provoked the world's current largest humanitarian displacement: since February 2022, one-third of Ukrainians have been forced to leave their homes, resulting in upwards of 7 million internally displaced persons. Estimates suggest that 60% of Ukraine's displaced persons are women, who face stressors including difficulty accessing necessary primary health and psychological care, restricted access to food and stable housing, and increased strain from separation from their social networks and additional family care responsibilities.

Early reports from Ukraine consistently describe the psychological distress that displaced women are presently experiencing. It is anticipated that nearly one in five people exposed to conflict will develop mental disorders, notably depressive and anxiety disorders. Thus, improving access to mental health prevention programs that mitigate development of mental disorders for women in Ukraine is critical.

This study will adapt a community-based Acceptance and Commitment Therapy (ACT) intervention to prevent the development symptoms of depression and anxiety among women displaced by war in Ukraine. ACT is an evidence-based approach that uses acceptance, mindfulness and behavioral change processes to improve psychological flexibility. Recently displaced women who screen positive for symptoms of depression and anxiety will be recruited. The investigators plan to adapt and evaluate a single-session ACT group intervention to limit effects of mental health distress among these displaced women.

The central hypothesis of this research is that an ACT-based intervention delivered in a humanitarian context will help displaced women in Ukraine learn skills to improve psychological flexibility, thereby decreasing symptoms of depression and anxiety and ultimately mitigating onset of mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Identify as a displaced woman within one year of migration
* Endorsing mild to moderate depressive symptoms (subscale score between 3 and 7) and/or anxiety symptoms (subscale score between 2 and 6) on the Mental Health Assessment Inventory (MHAI) but not exceeding the maximum score for either subscale (i.e., not exceeding 7 on the depressive symptoms subscale and not exceeding 6 on the anxiety symptoms subscale)
* Ability to provide informed consent
* Speak Ukrainian or Russian

Exclusion Criteria:

* Diagnosis of a depressive or anxiety disorder, or symptoms necessitating urgent referral for evaluation of suicidal or homicidal ideation
* Receipt of psychiatric care for depression or anxiety in the past 5 years
* A severe medical problem that inhibits ability to participate in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 120 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms | Baseline, 3 months
  Anxiety symptoms will be assessed using the Mental Health Assessment Inventory (MHAI) anxiety subscore which has 4 items, and each item is rated on a 3-point Likert scale where "0" means "none of the time" and "3" means "almost all of the time." Total score on the subscale ranges from 0-12 with higher scores indicating greater symptoms of anxiety.
Depressive symptoms | Baseline, 3 months
  Depressive symptoms will be assessed using the Mental Health Assessment Inventory (MHAI) depression subscore which has 6 items, and each item is rated on a 3-point Likert scale where "0" means "none of the time" and "3" means "almost all of the time." Total score on the subscale ranges from 0-36 with higher scores indicating greater symptoms of depression.

SECONDARY OUTCOMES:
Experiential avoidance | Baseline, 3-months
  Experiential avoidance will be assessed with the Multidimensional Experiential Avoidance Questionnaire (MEAQ) which is scored by summing up responses across its 62 items. Each item is rated on a 6-point Likert scale ranging from "strongly disagree" to "strongly agree". Higher scores indicate greater levels of experiential avoidance.
Psychological flexibility | Baseline, 3 months
  Psychological flexibility will be assessed using the Acceptance and Actions Questionnaire (AAQ-2) which has 7 items, and each item is rated on a 7-point Likert scale where "1" means "never true" and "7" means "always true". Scores can range from 7 to 49. The higher the score, the more someone tends to avoid unwanted thoughts and feelings, signifying less psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Lunze, MD DrPH MPH, Principal Investigator — CABUSchool of Medicine, General Internal Medicine
Locations (1):
- Alliance for Public Health, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT06679114/ICF_000.pdf